CLINICAL TRIAL: NCT00124904
Title: Biofeedback for Fecal Incontinence and Constipation
Brief Title: Biofeedback for Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RO1 DK57048a (completed); R01DK057048 (NIH)
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Fecal Incontinence
Keywords: Biofeedback; Incontinence
MeSH Terms: conditions — Fecal Incontinence | interventions — Biofeedback, Psychology

INTERVENTIONS:
Behavioral: Biofeedback
Behavioral: Kegel exercises

SUMMARY:
Fecal incontinence affects 2% of adults in the United States. Biofeedback has been recommended for the treatment of fecal incontinence because uncontrolled studies over the past 25 years suggest that these treatments are as effective as medical or surgical management and involve no risk. However, placebo-controlled trials are still lacking.

The aims of this study are: (1) to compare biofeedback to alternative therapies for which patients have a similar expectation of benefit; (2) to identify which patients are most likely to benefit; and (3) to assess the impact of treatment on quality of life.

DETAILED DESCRIPTION:
Study I is a long-term, prospective, single-blind study comparing biofeedback for fecal incontinence to a standard therapy (Kegel exercises) that is associated with a similar expectation of improvement (i.e., comparable placebo effect). Prior to randomization, patients will receive medical therapy (antidiarrheal medications as appropriate) and education for 4 weeks, and only patients who remain incontinent will be randomized. Anal canal squeeze pressures and rectal sensory thresholds will be tested before and after treatment. Patients will keep a diary throughout baseline and treatment, and they will be re-assessed at 3, 6, and 12 months. Treatment will consist of 6 clinic visits at 2-week intervals. The primary outcome is the patient's response to the question, "Have you had satisfactory relief of fecal incontinence (yes/no)?" This question is asked at 3 months following the end of treatment and at each follow-up visit. The investigators will develop a detailed treatment manual for fecal incontinence which would permit other investigators to replicate our study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 16 or above who have an average of one or more episodes of fecal incontinence per week

Exclusion Criteria:

* Previous biofeedback treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165
Dates: Start 1999-09; Study Completion 2006-12

PRIMARY OUTCOMES:
Proportion of subjects reporting adequate relief per treatment group

SECONDARY OUTCOMES:
Demonstrate association of improvement in quality of life with treatment outcome
Identify predictors of successful treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Department of Medicine, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Palsson OS, Heymen S, Whitehead WE. Biofeedback treatment for functional anorectal disorders: a comprehensive efficacy review. Appl Psychophysiol Biofeedback. 2004 Sep;29(3):153-74. doi: 10.1023/b:apbi.0000039055.18609.64. PMID 15497616
- [Background] Heymen S. Psychological and cognitive variables affecting treatment outcomes for urinary and fecal incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S146-51. doi: 10.1053/j.gastro.2003.10.040. PMID 14978652
- [Background] Jones KR, Heymen S, Whitehead WE. Biofeedback for Anorectal Disorders. In: Drutz HP, Herschorn S, Diamant NE (Eds), Female Pelvic Medicine and Reconstructive Pelvic Surgery. London, Springer-Verlag, 2003. Pp 313-325.
- [Background] Whitehead WE, Heymen S, Schuster MM. Motility as a therapeutic modality: biofeedback treatment of gastrointestinal disorders. Chapter 27. In MM Schuster, MD Crowell, KL Koch (Eds.), Schuster Atlas of Gastrointestinal Motility in Health and Disease. London, BC Decker Inc. 2002; 381-397.
- [Background] Heymen S, Jones KR, Ringel Y, Scarlett Y, Whitehead WE. Biofeedback treatment of fecal incontinence: a critical review. Dis Colon Rectum. 2001 May;44(5):728-36. doi: 10.1007/BF02234575. PMID 11357037
- [Background] Heymen S, Jones KR, Ringel Y, Scarlett Y, Drossman D, Whitehead WE (abstract). Biofeedback for fecal incontinence and constipation: the role of medical management and education. Gastro 2001 (suppl 1):120, A397.
- [Result] Scarlett Y. Medical management of fecal incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S55-63. doi: 10.1053/j.gastro.2003.10.007. PMID 14978639
- [Result] Heymen S, Scarlett Y, Whitehead WE. Education and medical management resolve fecal incontinence in 35%, but depression and greater symptom severity predict a poor response. Am J Gastroenterol Suppl 2004;99:T1374.
- [Result] Heymen S, Scarlett Y, and Whitehead WE. Elevated Beck Depression Inventory (BDI) Scores Predict Biofeedback Treatment Failure for Fecal Incontinence and Constipation (abstract). Gastroenterology 2003,124:4(suppl 1)A-685.
- [Derived] Vonthein R, Heimerl T, Schwandner T, Ziegler A. Electrical stimulation and biofeedback for the treatment of fecal incontinence: a systematic review. Int J Colorectal Dis. 2013 Nov;28(11):1567-77. doi: 10.1007/s00384-013-1739-0. Epub 2013 Jul 31. PMID 23900652
- See also: Center website — http://www.med.unc.edu/ibs